CLINICAL TRIAL: NCT05265884
Title: Effect of Kinesiotaping on Myofascial Pain Syndrome Post Neck Dissection Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moshira Medhat Mahmoud Esmail, Moshira Medhat ,Assistant lecturer of physical therapy,cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003435
Record Dates: First submitted 2022-01-15; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Myofascial Pain Syndrome
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Kinesio taping group)(Experimental group): (Experimental): This group includes 30 patients who will receive Kinesiotaping, in additional to traditional treatment (ROM exercises, stretching exercises, and Deep friction message) 3 times per week for one month.
  Interventions: Device: Kinesiotaping; Behavioral: traditional therapy intervention
- Group B (control group) (Active Comparator): This group includes 30 patients who will receive traditional treatment only (ROM exercises, stretching exercises, and Deep friction message) 3 times per week for 1 month.
  Interventions: Behavioral: traditional therapy intervention

INTERVENTIONS:
Device: Kinesiotaping — The tape is waterproof, porous, and adhesive. The width is 5 cm and thickness of 0.5 mm will be used in this study. This tape is with elastic core wrapped within cotton and capable of stretching up to 140-150%, applies heat-sensitive acrylic adhesive to avoid risk of latex allergy .The tape without medicinal properties is water resistant and can remain on the skin for 3 to 5 days. It will be applied two times per week for one month
  Arms: Group A (Kinesio taping group)(Experimental group):
Behavioral: traditional therapy intervention — traditional treatment (ROM exercises, stretching exercises, and Deep friction message) 3 times per week for one month.

SUMMARY:
The purpose of the study is to evaluate the effect of Kinesio taping on myofascial pain syndrome post neck dissection surgery.

DETAILED DESCRIPTION:
In this part of the study, the materials and methods will be presented under the following headings: subjects, equipment, procedures of the study and the statistical procedures.

1. Subjects:

   Sixty patients from both genders who have cervical myofascial pain syndrome (MPS) following a neck dissection surgery will participate in this study. Their ages will be ranged from 30 to 45 years. The participants will be selected from the National Cancer Institute, Cairo University and randomly distributed into two equal groups.

   1.1 Design of the study:

   In this study the patients will be randomly assigned into two equal groups (30 patients for each group):

   1.1(a) Group A (Kinesio taping group): This group includes 30 patients who will receive Kinesiotaping, in additional to traditional treatment (ROM exercises, stretching exercises, and Deep friction message) 3 times per week for one month.

   1.1(b) Group B This group includes 30 patients who will receive traditional treatment only (ROM exercises, stretching exercises, and Deep friction message) 3 times per week for 1 month.
2. Equipment:

2.1- Measurement equipment: 2.1.a-Visual analogue scale (VAS): The Visual analogue Scale (VAS) has been in use for the measurement of intangible quantities such as pain, quality of life and anxiety since the 1920s. It consists of a line usually 100 mm in length, with anchor descriptors such as (in the pain context) "no pain" and "worst pain imaginable". The patient makes a mark reflecting his or her perception, and the distance from the left endpoint to the mark is measured, in mm. The VAS was initially used in psychology for the measurement of mood disorders, and was used for the measurement of pain from the mid-1960s .

2.1.b- A pressure algometer: - A pressure algometer will be used for pressure pain threshold (PPT) assessment on the trigger spots. It contains a rubber disk (1 cm2surface), attached to a pressure pole and inserted into a gauge, for recording the pressure in kilograms .

2.1.C-Goniometer: The term goniometry is derived from two Greek words, gonia, meaning "angle" and metron, meaning "measurement". Goniometer has different types; the most used is the universal standard goniometer, which is either made with plastic or metal tool. It consists of a stationary arm, a movable arm, and a fulcrum. By aligning this with the axis of a joint, the degree of motion can be measured in a single plane .

-The active ROM of neck joint (lateral flexion and rotation on both sides.) will be measured using a universal standard goniometer when the patient is in sitting position.

2.2-Therapeutic equipment and tools:

Kinesio tape:

The tape (Kinesio Tex Tape; Kinesio Holding Corporation, Albuquerque, NM) is waterproof, porous, and adhesive. The width is 5 cm and thickness of 0.5 mm will be used in this study. This tape is with elastic core wrapped within cotton and capable of stretching up to 140-150%, applies heat-sensitive acrylic adhesive to avoid risk of latex allergy .The tape without medicinal properties is water resistant and can remain on the skin for 3 to 5 days. It will be applied two times per week for one month.

ELIGIBILITY:
Inclusion Criteria:

* Both genders with age range between 30 to 45 years will participate in this study.
* A history of MPS involving upper trapezius for at least 3 months.
* Moderate to severe pain (VAS score >4).

Exclusion Criteria:

* The potential participants will be excluded if they meet one of the following criteria:

  * A wound in the affected area
  * A cervical disk lesion
  * Myelopathy or radiculopathy
  * Cervical spine fracture or spondylolisthesis
  * Rheumatoid arthritis,
  * Epilepsy or any psychological disorders

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
assessing and quantifying pain exhibited by the patients | 1 month
  Visual analogue scale (VAS):
  The Visual analogue Scale (VAS) has been in use for the measurement of intangible quantities such as pain, quality of life and anxiety since the 1920s. It consists of a line usually 100 mm in length, with anchor descriptors such as (in the pain context) "no pain" and "worst pain imaginable". The patient makes a mark reflecting his or her perception, and the distance from the left endpoint to the mark is measured, in mm. The VAS was initially used in psychology for the measurement of mood disorders, and was used for the measurement of pain from the mid-1960s The VAS will be used for assessing and quantifying pain exhibited by the patients through a 0-10 scale. Each subject twill be informed to mark the line according to the pain intensity experienced at that particular time where 0 means no pain and 10 means worst conceivable pain

SECONDARY OUTCOMES:
pressure pain threshold (PPT) | 1 month
  A pressure algometer:
  Pressure algometer(Somedic AB, Farsta, Sweden)will be used for pressure pain threshold (PPT) assessment on the trigger spots. Participants will be informed to elucidate when the pressure sensation became painful and to immediately release the pressure. The most painful point will be marked by a waterproof marker on the initial visit. The average of three measurements will be recorded

OTHER OUTCOMES:
Range of motion | 1 month
  Neck ROM will be measured using the universal standard goniometer while patients in sitting position to remove errors and movement compensation. The subjects will be asked for sitting with their back straight and strapped to the back of the chair. Subject's ankles, knees and hips will be positioned at right angle and arms will be folded across the chest to minimize thoracic movement. The active ROM of the neck (lateral flexion and rotation on both sides.) will be measured using the universal standard goniometer when the patient is in sitting position.

CONTACTS AND LOCATIONS:
Overall Officials: faculty of physical therapy, Study Director — teaching assistant at faculty of physical therapy Cairo university
Locations (1):
- Faculty Of phyical tehrapy, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No